CLINICAL TRIAL: NCT00428220
Title: An Open-label Sunitinib Malate (su011248) Continuation Protocol For Patients Who Have Completed A Prior Sunitinib Study And Are Judged By The Investigator To Have The Potential To Benefit From Sunitinib Treatment
Brief Title: A Continuation Study Using Sunitinib Malate For Patients Leaving Treatment On A Previous Sunitinib Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181114; 2006-006538-16 (EudraCT Number)
Record Dates: First submitted 2007-01-26; First posted 2007-01-29 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Metastatic Breast Cancer; Advanced Breast Cancer; Metastatic Castration Resistant Prostate Cancer; Metastatic Renal Cell Cancer; Non-Small Cell Lung Cancer; Thyroid Cancer; Advanced/Metastatic Non-Small Cell Lung Cancer; Advanced Gastric Cancer; Gastrointestinal Stromal Tumor; Hepatocellular Carcinoma; Pancreatic Islet Cell Carcinoma; Pancreatic Neuroendocrine Tumor
Keywords: Potentially other tumor types in the future
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Thyroid Neoplasms; Gastrointestinal Stromal Tumors; Carcinoma, Hepatocellular; Somatostatinoma; Adenoma, Islet Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Sunitinib will be administered in a continuous daily dose (oral, once per day). Starting dose will be 37.5 mg daily unless the patient was on a different dose (25 mg or 50 mg daily) on the previous trial. In that case, they will begin treatment on this study at the same dose used at the end of the previous study.
  The protocol now allows for patients on dosing regimens other than only continuous dosing (e.g. 4/2, etc.) to be enrolled if eligible.
  Interventions: Drug: sunitinib

INTERVENTIONS:
Drug: sunitinib — sunitinib

SUMMARY:
This is a study using sunitinib for patients ending treatment on a previous sunitinib malate protocol to continue to receive sunitinib. The patient must have been enrolled in one of the following studies: A6181030, A6181064, A6181078, A6181087, A6181094, A6181107, A6181108, A6181110, A6181111, A6181112, A6181113, A6181120, A6181126 and A6181170. Other Pfizer sponsored sunitinib studies may be included in the future.

ELIGIBILITY:
Inclusion Criteria:

* Must have ended treatment from one of the following sunitinib studies: A6181030, A6181064, A6181078, A6181087, A6181094, A6181107, A6181108, A6181110, A6181111, A6181112, A6181113, A6181120, A6181126 and A6181170. Other Pfizer sponsored sunitinib studies may be included in the future.

Exclusion Criteria:

* See inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2007-07; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (112):
- United States (14):
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - Investigational Drug Service, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Siteman Cancer Center, City of Saint Peters, Missouri
  - Siteman Cancer Center-West County, Creve Coeur, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, Siteman Cancer Center, St Louis, Missouri
  - Comprehensive Cancer Center of Nevada, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - US Oncology Research and Clinical Pharmacy (Drug Shipment Only), Fort Worth, Texas
  - The Strelitz Diabetes Institute of Eastern Virginia Medical School, Norfolk, Virginia
- Argentina (4):
  - Instituto Oncologico de Cordoba, Nueva Cordoba, Nueva Cordoba
  - Clinica Viedma, Viedma, Río Negro Province
  - Centro Oncológico Rosario, Rosario, Santa Fe Province
  - Centro Medico San Roque, San Miguel de Tucumán
- Australia (5):
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Department of Medical Oncology, Adelaide, South Australia
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Mount Medical Centre, Perth, Western Australia
- Belgium (7):
  - Hopital Erasme / Gastroenterologie, Brussels
  - Cliniques Universitaires Saint Luc / Gastroentérologie, Brussels
  - Cliniques Universitaires Saint-Luc, Oncologie, Brussels
  - UZ Gasthuisberg, Department Internal Medicine - Gastroenterology - Gastro-intestinal Oncology, Leuven
  - Centre Hospitalier Universitaire de Liege, Liège
  - Algemeen Ziekenhuis Nikolaas, Sint-Niklaas
  - AZ Sint-Augustinus, Oncologisch Centrum, Wilrijk
- Brazil (4):
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Centro de Oncologia do Instituto de Radiologia, São Paulo, São Paulo
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo, São Paulo
- Canada (8):
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - QEII Health Sciences Centre - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - QEII Health Sciences Centre - Victoria General Site, Halifax, Nova Scotia
  - QEII Health Sciences Centre - Halifax Infirmary Site, Halifax, Nova Scotia
  - London Regional Cancer Program, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUM, Hopital Saint-Luc, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
- Colombia (3):
  - Fundacion Centro de Investigacion Clinica CIC, Medellín, Anquioquia
  - Hospital Universitario San Vicente de Paul, Medellín, Antioquia
  - Clinica Astorga, Medellín, Antioquia
- France (14):
  - Centre Antoine Lacassagne, Nice, Cedex 02
  - Hopital Beaujon, Clichy, Cedex
  - Groupe Hospitalier Cochin, Cancer Quest AP-HP, Paris, Cedex
  - CHU-Hôpital Jean Minjoz, Besançon
  - Hopital Saint-Andre, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Polyclinique du Bois, Lille
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital Edouard Herriot, Lyon
  - Chu La Timone, Marseille
  - Clinique Hartmann, Neuilly-sur-Seine
  - Hopital Saint-Antoine, Paris
  - Centre Eugene Marquis, Rennes
- Germany (9):
  - Klinik fuer Innere Medizin, Gastroenterologie, Onkologie, Endokrinologie, Bad Berka
  - Universitaetsklinikum Charité, Campus Virchow Klinikum, Berlin
  - eps - early phase GmbH, Jena
  - Frauenaerzte Pruener Gang, Kiel
  - Klinik fuer Frauenheilkunde und Geburtshilfe, Universitaetsklinikum Schleswig-Holstein, Lübeck
  - Universitaetsklinikum Schleswig-Holstein, Campus Luebeck, Lübeck
  - Universitaetsklinikum Giessen und Marburg, Standort Marburg, Marburg
  - Rhoen Klinikum Meiningen, Gynaekologie und Geburtshilfe, Meiningen
  - Frauenklinik und Poliklinik, Klinikum rechts der Isar, Technische Universitaet Muenchen, München
- Hong Kong (6):
  - Department of Clinical Oncology, Tuen Mun Hospital, Tuenmen, New Territories
  - Queen Mary Hospital, Hong Kong
  - Division of Haematology/Oncology, Department of Medicine, Queen Mary Hospital,, Hong Kong
  - Queen Elizabeth Hospital, Department of Clinical Oncology, Kowloon
  - Tuen Mun Hospital, Department of Clinical Oncology, Tuen Mun, New Territories
  - UNIMED Medical Institute, Wan Chai
- Mexico (2):
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez Centro Universitario contra el cancer, Monterrey, Nuevo León
  - Hospital Christus Muguerza del Parque, Chihuahua City
- Cancer Care Clinic, Quezon City, Metro Manila, Philippines
- Singapore (2):
  - National University Hospital/Department of Heamatology-Oncology, Singapore
  - National Cancer Center/Department of Medical Oncology, Singapore
- South Korea (6):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital / Department of Internal Medecine, Seoul, Republic of Korea
  - Asan Medical Center, Division of Oncology, Department of Internal Medicine, Seoul, Republic of Korea
  - Yeungnam University Medical Center/Department of Internal medicine, Daegu
  - Severance Hospital, Yonsei Cancer Center, Yonsei University College of Medicine, Seoul
- Spain (8):
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Fundacion Hospital Alcorcon, Alcorcón, Madrid
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Servicio de Oncologia, Barcelona
  - Centro Oncologico Md Anderson International España, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
- Taiwan (9):
  - Chi Mei Medical Center, Liouying, Liouying Township, Tainan,, Taiwan
  - Chi-Mei Medical Center, YungKang City, Tainan, Taiwan
  - Chang Gung Medical Foundation, Linkou Branch, Guishanli, Taoyuan
  - Changhua Christian Hospital, Changhua
  - Chung-Ho Memorial Hospital, Kaohsiung Medical University/Department of Surgery, Kaohsiung City
  - Taichung Veterans General Hospital, Department of Surgery, Taichung
  - National Taiwan University Hospital/Department of Oncology, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Div. of Hematology/Oncology, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (10):
  - Division of Surgery and Oncology, Liverpool, Merseyside
  - Deparment of Cardiology, Glasgow
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - Dainton Building, Leeds
  - St James' Institute of Oncology, Leeds
  - Management Offices, 4th Floor, Thomas Guy House, London
  - Royal Marsden Hospital, London
  - Department of Medical Oncology, Manchester
  - Cardiology Department, Wythenshawe Hospital, Manchester
  - Nottingham City Hospital, Nottingham

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181114&StudyName=A%20Continuation%20Study%20Using%20Sunitinib%20Malate%20For%20Patients%20Leaving%20Treatment%20On%20A%20Previous%20Sunitinib%20Study.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this open-label extension study, access to sunitinib was provided to participants who had participated in a previous parent study and who had been judged by the Investigator to have likely clinical benefit from continuing sunitinib dosing.
Pre-assignment Details: Participants receiving sunitinib in previous studies began treatment in this study with the last dose they were taking in the parent or extension study. Participants were to continue to access sunitinib on this protocol as long as there was evidence of disease control and/or clinical benefit in the judgment of the Investigator.
Groups:
- Sunitinib: Participants receiving treatment on single-agent sunitinib on continuous dosing regimens returned for study visits at Day 28, and every 8 weeks thereafter. Participants on regimens other than single-agent sunitinib on continuous dosing followed the schedule of activities from their parent or extension protocol. Sunitinib-naïve participants (ie, those not treated with sunitinib in the previous parent study) received a starting dose of 37.5 mg sunitinib once daily.
Period: Overall Study
Arm/Group | Sunitinib
Started | 223
Completed | 0
Not Completed | 223
Not completed — Participant died | 8
Not completed — Global deterioration of health status | 7
Not completed — Lost to Follow-up | 4
Not completed — Objective progression or relapse | 123
Not completed — Participant refused continued treatment | 7
Not completed — Adverse Event | 51
Not completed — Other | 23

BASELINE CHARACTERISTICS:
Population: The safety population was defined as all participants enrolled in the study who received at least one dose of study drug in this study.
Arm/Group | Sunitinib
Number analyzed (Participants) | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130
  Male | 93

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) (All Causalities)
Description: Assessment of AEs included type, incidence, severity (graded by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], Version 3.0, timing, seriousness, and relatedness; and laboratory abnormalities.
Time Frame: From first day of treatment on the current study up to 28 days post the last dose of study treatment
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 223
participants
  Participants with adverse events (AE) | 221
  Participants with serious adverse events (SAE) | 90
  Participants with grade 3 or 4 AEs | 174
  Participants with grade 5 AEs | 24
  Participants discontinued due to AEs | 67
  Participants with dose reduction due to AEs | 66
  Temporary discontinuations due to AEs | 146

2. Primary Outcome: Number of Participants With Treatment-emergent AEs (Treatment-Related)
Description: as for outcome 1
Time Frame: From first day of treatment on the current study up to 28 days post the last dose of study treatment
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 223
participants
  Participants with AE | 217
  Participants with SAE | 39
  Participants with grade 3 or 4 AEs | 146
  Participants with grade 5 AEs | 0
  Participants discontinued due to AEs | 29
  Participants with dose reduction due to AEs | 64
  Temporary discontinuations due to AEs | 135

3. Other Pre Specified Outcome: Summary of Duration of Clinical Benefit
Description: Duration of clinical benefit is defined as the length of time participants remain on sunitinib from the first day of treatment on the parent protocol until the end of sunitinib treatment in this study (A6181114). For participants who were on placebo or a comparator drug in the parent study, duration of clinical benefit is defined as the length of time participants are on sunitinib in this study.
Time Frame: From the first day of treatment in parent study until last day of treatment in A6181114 study.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Weeks
Groups:
- Sunitinib 1: Parent Study: A6181078
- Sunitinib 2: Parent Study: A6181087
- Sunitinib 3: Parent Study: A6181094
- Sunitinib 4: Parent Study: A6181107
- Sunitinib 5: Parent Study: A6181110
- Sunitinib 6: Parent Study: A6181111
- Sunitinib 7: Parent Study: A6181112
- Sunitinib 8: Parent Study: A6181113
- Sunitinib 9: Parent Study: A6181120
- Sunitinib 10: Parent Study: A6181126
- Sunitinib 11: Parent Study: A6181170
Arm/Group | Sunitinib 1 | Sunitinib 2 | Sunitinib 3 | Sunitinib 4 | Sunitinib 5 | Sunitinib 6 | Sunitinib 7 | Sunitinib 8 | Sunitinib 9 | Sunitinib 10 | Sunitinib 11
Number analyzed (Participants) | 3 | 1 | 2 | 69 | 38 | 95 | 8 | 1 | 3 | 1 | 2
Weeks | 186.6 (68.2) | 76.0 (NA) — Only one datum, hence no standard deviation. | 157.5 (6.2) | 22.1 (25.2) | 122.9 (73.4) | 76.6 (69.0) | 71.6 (26.2) | 198.9 (NA) — Only one datum, hence no standard deviation. | 142.2 (23.6) | 183.6 (NA) — Only one datum, hence no standard deviation. | 227.5 (57.9)

ADVERSE EVENTS:
Time Frame: From first day of treatment on the current study up to 28 days post the last dose of study treatment
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 90/223
Other Adverse Events (participants affected / at risk) | 219/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=223)
Anaemia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Abdominal adhesions (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 8
Abdominal pain upper (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 6
Duodenitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Haematemesis (Gastrointestinal disorders) | 2
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Mallory-weiss syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Peritoneal haemorrhage (Gastrointestinal disorders) | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 3
Chest pain (General disorders) | 2
Disease progression (General disorders) | 12
Fatigue (General disorders) | 1
Gait disturbance (General disorders) | 1
General physical health deterioration (General disorders) | 5
Generalised oedema (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Oedema (General disorders) | 1
Pyrexia (General disorders) | 5
Sudden death (General disorders) | 1
Biliary colic (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 2
Hepatic failure (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lymphangitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pneumonia bacterial (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Blood calcium increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Urosepsis (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Scrotal erythema (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Aortic dissection (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Pelvic venous thrombosis (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
Lipase increased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=223)
Anaemia (Blood and lymphatic system disorders) | 41
Leukopenia (Blood and lymphatic system disorders) | 35
Neutropenia (Blood and lymphatic system disorders) | 76
Thrombocytopenia (Blood and lymphatic system disorders) | 57
Hypothyroidism (Endocrine disorders) | 24
Lacrimation increased (Eye disorders) | 13
Abdominal distention (Gastrointestinal disorders) | 20
Abdominal pain (Gastrointestinal disorders) | 62
Abdominal pain upper (Gastrointestinal disorders) | 46
Constipation (Gastrointestinal disorders) | 41
Diarrhoea (Gastrointestinal disorders) | 142
Dry mouth (Gastrointestinal disorders) | 14
Dyspepsia (Gastrointestinal disorders) | 36
Gastritis (Gastrointestinal disorders) | 13
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 14
Haemorrhoids (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 77
Stomatitis (Gastrointestinal disorders) | 39
Vomiting (Gastrointestinal disorders) | 61
Asthenia (General disorders) | 67
Chest pain (General disorders) | 14
Face oedema (General disorders) | 17
Fatigue (General disorders) | 83
Mucosal inflammation (General disorders) | 58
Oedema peripheral (General disorders) | 30
Pain (General disorders) | 13
Pyrexia (General disorders) | 26
Gingivitis (Infections and infestations) | 12
Nasopharyngitis (Infections and infestations) | 18
Upper respiratory tract infection (Infections and infestations) | 17
Alanine aminotransferase increased (Investigations) | 21
Aspartate aminotransferase increased (Investigations) | 15
Blood creatinine increased (Investigations) | 13
Haemoglobin decreased (Investigations) | 20
Neutrophil count decreased (Investigations) | 16
Platelet count decreased (Investigations) | 19
Weight decreased (Investigations) | 36
Decreased appetite (Metabolism and nutrition disorders) | 76
Hyperglycaemia (Metabolism and nutrition disorders) | 13
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 31
Back pain (Musculoskeletal and connective tissue disorders) | 47
Bone pain (Musculoskeletal and connective tissue disorders) | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 18
Myalgia (Musculoskeletal and connective tissue disorders) | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 36
Dizziness (Nervous system disorders) | 16
Dysgeusia (Nervous system disorders) | 60
Depression (Psychiatric disorders) | 14
Insomnia (Psychiatric disorders) | 35
Cough (Respiratory, thoracic and mediastinal disorders) | 35
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 43
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14
Alopecia (Skin and subcutaneous tissue disorders) | 17
Dry skin (Skin and subcutaneous tissue disorders) | 21
Erythema (Skin and subcutaneous tissue disorders) | 19
Hair colour changes (Skin and subcutaneous tissue disorders) | 55
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 13
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 83
Headache (Nervous system disorders) | 44
Rash (Skin and subcutaneous tissue disorders) | 30
Skin discolouration (Skin and subcutaneous tissue disorders) | 26
Yellow skin (Skin and subcutaneous tissue disorders) | 22
Hypertension (Vascular disorders) | 64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.